CLINICAL TRIAL: NCT06557200
Title: Empowering Early Parenthood: A Digital Psychoeducational Support Intervention for Postnatal Well-being
Brief Title: A Virtual Support Intervention for Postnatal Well-being
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Putra Malaysia (Other)
Collaborators: University of Lahore (Other)
Responsible Party: Principal Investigator, Arshed Muhammad, PhD studentship, Universiti Putra Malaysia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: UIPT
Record Dates: First submitted 2024-08-13; First posted 2024-08-16 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Postnatal Depression; Mother-Infant Interaction
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Intervention Model Description: A virtual and in-person, personal and group-based intervention will be delivered-educational information on infant behavior and changes in interpersonal dynamics associated with parenting. Modules aimed at understanding and managing infant behavior include information on infant temperament. Personal support will be provided by face-to-face education and WhatsApp messages and videos. Group support will be provided by mothers and their partners or a support person group discussion.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Participants, Care providers, and outcome assessors will be blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): A virtual and in-person, personal and group-based intervention will be delivered-educational information on infant behavior and changes in interpersonal dynamics associated with parenting. Modules aimed at understanding and managing infant behavior include information on infant temperament. Personal support will be provided by face-to-face education and WhatsApp messages and videos. Group support will be provided by mothers and their partners or a support person group discussion.
  Interventions: Behavioral: Digital Infant- parents support
- Control (No Intervention): No intervention will be provided except usual care

INTERVENTIONS:
Behavioral: Digital Infant- parents support — A virtual and in-person, personal and group-based intervention will be delivered-educational information on infant behavior and changes in interpersonal dynamics associated with parenting. Modules aimed at understanding and managing infant behavior include information on infant temperament. Personal support will be provided by face-to-face education and WhatsApp messages and videos. Group support will be provided by mothers and their partners or a support person group discussion.
  Arms: Intervention group

SUMMARY:
Postnatal depression (PND) and anxiety are significant public health concerns affecting a substantial proportion of new mothers worldwide. These conditions can have profound consequences for both maternal and infant well-being, including increased risk of

1. maternal morbidity
2. impaired parent-infant bonding
3. long-term developmental challenges for the child.

DETAILED DESCRIPTION:
Despite the prevalence and impact of PND and anxiety, access to timely and effective mental health care for postpartum women remains limited, particularly in resource-constrained settings.

Limited Research: There has been a historical underinvestment in mental health research in Pakistan, especially in maternal mental health.

Cultural Stigma: Mental health issues, particularly postpartum depression, are often stigmatized, leading to underreporting.

Data Infrastructure: Robust data collection and analysis systems for mental health are still developing in Pakistan The rationale for this study is grounded in the significant public health burden imposed by postnatal depression (PND) and anxiety, coupled with the limitations of traditional care models. Despite advancements in maternal and child health, postpartum mental health remains a neglected area in many countries, including Pakistan.

ELIGIBILITY:
Inclusion Criteria:

* Pakistani female aged 18-45 years
* Recent childbirth (within 0-6 weeks)
* Access to a smartphone or computer with internet connectivity
* Able to understand and communicate in Urdu or English
* Willing to provide informed consent

Exclusion Criteria:

* Pre-existing severe mental illness (e.g., schizophrenia, bipolar disorder)
* Current substance abuse or dependence
* Limited or no access to the internet or smartphone
* Inability to understand or communicate in Urdu or English
* Pregnancy complications requiring intensive care
* Infants with severe medical conditions requiring hospitalization

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1400 (Estimated)
Dates: Start 2024-08-15 (Estimated); Primary Completion 2025-07-15 (Estimated); Study Completion 2025-08-10 (Estimated)

PRIMARY OUTCOMES:
Post natal depression | Post natal Depression measured at baseline and 12 months
  Edinburgh Postnatal Depression Scale (EPDS): A standardized self-report questionnaire to assess symptoms of postnatal depression. Scores are between 0 and 30, with scores 13 and above indicating depressive illness, or a high risk of developing a depressive disorder. Scores of 13 indicate an 80% chance that the mother has depression.
Post natal anxiety | Post natal Anxiety measured at baseline and 12 months
  Generalized Anxiety Disorder-7 (GAD-7): A self-report measure to assess symptoms of generalized anxiety disorder. The GAD-7 scores were also represented with clinical categorizations of anxiety levels as follows: GAD-7 score of 0-4 (none), 5-9 (mild), 10-14 (moderate), and 15-21 (severe).
Intervention usage | Intervention usage measured at 12 months
  Intervention usage will be assessed by tracking participants' engagement with the online platform, including login frequency, module completion, and time spent on the platform.

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmad Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
Study protocol, Statistical plan, Results will be desseminated through publications

REFERENCES:
- [Background] Woody CA, Ferrari AJ, Siskind DJ, Whiteford HA, Harris MG. A systematic review and meta-regression of the prevalence and incidence of perinatal depression. J Affect Disord. 2017 Sep;219:86-92. doi: 10.1016/j.jad.2017.05.003. Epub 2017 May 8. PMID 28531848
- [Background] Hahn-Holbrook J, Cornwell-Hinrichs T, Anaya I. Economic and Health Predictors of National Postpartum Depression Prevalence: A Systematic Review, Meta-analysis, and Meta-Regression of 291 Studies from 56 Countries. Front Psychiatry. 2018 Feb 1;8:248. doi: 10.3389/fpsyt.2017.00248. eCollection 2017. PMID 29449816
- [Background] Coo S, Garcia MI, Mira A, Valdes V. The Role of Perinatal Anxiety and Depression in Breastfeeding Practices. Breastfeed Med. 2020 Aug;15(8):495-500. doi: 10.1089/bfm.2020.0091. Epub 2020 Jun 9. PMID 32522015
- [Background] Rojas G. Análisis de La Situación de Uso de Servicios y Acceso a Tratamiento de La Depresión Posparto En Centros APS de La Región Metropolitana. Santiago, Chile: Universidad de Chile, http://www.crececontigo.gob.cl/wp-content/uploads/2015/11/5-Informe-Final-Analisis-de-lasituacion-de-uso-de-servicio-y-acceso-a-tratamiento-de-la-depresion-posparto.pdf (2013, accessed 15 January 2022).
- [Background] Priel A, Djalovski A, Zagoory-Sharon O, Feldman R. Maternal depression impacts child psychopathology across the first decade of life: Oxytocin and synchrony as markers of resilience. J Child Psychol Psychiatry. 2019 Jan;60(1):30-42. doi: 10.1111/jcpp.12880. Epub 2018 Feb 27. PMID 29484656